CLINICAL TRIAL: NCT04618523
Title: Efficacy and Safety of Artesunate-amodiaquine and Artemether-lumefantrine in the Treatment of Uncomplicated Plasmodium Falciparum Malaria in the Democratic Republic of the Congo: a Randomized Controlled Trial
Brief Title: Safety and Efficacy of Recommended Antimalarial in the Democratic Republic of the Congo
Acronym: TET2020
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ministry of Public Health, Democratic Republic of the Congo (Other Government)
Collaborators: University of Kinshasa (Other); World Health Organization (Other); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other)
Responsible Party: Principal Investigator, Prof. Gauthier Mesia Kahunu, Professor, Ministry of Public Health, Democratic Republic of the Congo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASAQ-LA 2019 DRC
Record Dates: First submitted 2020-10-22; First posted 2020-11-06 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artesunate-amodiaquine (Experimental): Tablets containing 25 mg of artesunate and 67.5 mg of amodiaquine: one tablet daily for three days for children weighing 4.5 to 8 kg, and tablets containing 50 mg of artesunate and 135 mg of amodiaquine: one tablet daily for three days for children weighing 9 to 17 kg.
  Interventions: Drug: Artesunate-amodiaquine
- Artemether-lumefantrine (Experimental): Tablets containing 20 mg of Artemether and 120 mg of Lumefantrine. Each dose to be taken with high-fat food or drinks (for example milk).
  One tablet twice daily for children weighing 5 to <15 kg, two tablets twice daily for those weighing 15 to <25 kg and three tablets twice daily for those weighing 25 to < 35 kg, for three days.
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Artesunate-amodiaquine — Artemisinin-based combination treatment
  Other Names: ASAQ Winthrop®
  Arms: Artesunate-amodiaquine
Drug: Artemether-lumefantrine — Artemisinin-based combination treatment
  Other Names: Coartem dispersible®
  Arms: Artemether-lumefantrine

SUMMARY:
Despite all efforts, malaria remains a public health concern, in particular in the Democratic Republic of the Congo (DRC). The National Malaria Control program recommends artemisinin-based combination treatments (ACTs), in particular artesunate-amodiaquine or artemether-lumefrantrine for the treatment of uncomplicated malaria. Previous studies indicated that ACTs are still effective, with efficacy above the required threshold of 90%. It is required to assess regularly the efficacy of antimalarial drugs. I In case of increasing failure rates, alternative options can be decided ontime.

The purpose of this trial is to assess efficacy and safety of artesunate-amodiaquine (ASAQ Winthrop®) and artemether-lumefantrine (Coartem Dispersible®) at day 28 in the treatment of uncomplicated Plasmodium falciparum malaria in six surveillance sites around DRC.

DETAILED DESCRIPTION:
This is a phase IV, randomized, open label, 2-arm trial. It will be performed in six malaria sentinel site around the Democratic Republic of the Congo. Children aged 6 to 59 months with confirmed Plasmodium falciparum uncomplicated malaria will be enrolled after informed consent granted by a parent or guardian. They will be randomized to receive either artesunate-amodiaquine or artemether lumefrantrine during 3 days (directly observed treatment) and then followed up until day 28. At each visit, clinical examination will be done and malaria testing as well. Hemoglobin level will be measured on recruitment day and then every two weeks until day 28.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6 to 59 months
* monoinfection with Plasmodium falciparum with asexual parasite count of 2,000 to 200,000/µL
* axillary temperature ≥ 37.5 °C
* ability to swallow oral medication
* ability and willingness to comply with the protocol for the duration of the study and to comply with the study visit schedule;
* informed consent from a parent or aguardian
* living within the study catchment area

Exclusion Criteria:

* presence of general danger signs in children aged under 5 years or signs of severe falciparum malaria according to the definitions of WHO;
* body weight < 5kg
* hemoglobin level < 5g/ dL or hematocrit < 15%
* presence of severe malnutrition
* presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* regular medication, which may interfere with antimalarial pharmacokinetics;
* malaria treatment within 2 days prior to recruitment
* history of hypersensitivity reactions or contraindications to any of the medicines being tested or used as alternative treatment

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1117 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
PCR adjusted efficacy | 28 days
  absence of fever and negative blood smear during the follow-up until day 28 and new infections occurred during the follow-up.

SECONDARY OUTCOMES:
Proportion of adverse events and serious adverse events | 28 days
  Number of adverse events and serious adverse events that every participant will experience
Proportion of participants with positive blood smear at day 3 | 3 days
  Number of participants who will still have parasites on day 3

OTHER OUTCOMES:
Presence of Plasmodium falciparum resistance markers and deletion of HRP2 | 28 days
  Resistance markers and deletion of HRP2 will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Gauthier Mesia Kahunu, PhD, Principal Investigator — University of Kinshasa
Locations (6):
- Democratic Republic of the Congo (6):
  - Centre Evangélique de Coopération, Kimpese, Bas-Congo Province
  - Centre de Santé Lupidi 1, Kapolowe, Haut-Katanga
  - Centre de Santé de Référence Mikalayi, Kazumba, Kasai-Central
  - Centre de Santé de Référence Rutshuru, Rutshuru, North Kivu
  - Centre de Santé Foyer Social, Kisangani, Tshopo
  - Centre de Santé Boende 2 Nsele, Boende, Tshuapa

IPD SHARING:
Plan to Share IPD: No